CLINICAL TRIAL: NCT06281665
Title: Treatment With Aspirin After Preeclampsia: TAP Trial
Acronym: TAP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Malamo Countouris (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Malamo Countouris, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STUDY23080099; K23HL168356 (NIH)
Record Dates: First submitted 2024-02-15; First posted 2024-02-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hypertensive Disorder of Pregnancy; Pre-Eclampsia; Hypertension; Eclampsia; Gestational Hypertension; Cardiovascular Diseases; Toxemia; Pregnancy Complications; Vascular Diseases; Hypertension, Pregnancy Induced; Hypertension;Pre-Eclamptic
Keywords: Hypertension
MeSH Terms: conditions — Toxemia; Pre-Eclampsia; Hypertension; Eclampsia; Hypertension, Pregnancy-Induced; Cardiovascular Diseases; Pregnancy Complications; Vascular Diseases | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: This is a pilot randomized, single-center, double-blind placebo-control study of low-dose aspirin in postpartum individuals with preeclampsia. Individuals will be randomized at the time of delivery 1:1 to 81mg of low-dose aspirin or similar-appearing placebo daily for six months postpartum. Treatment and control groups will monitor home blood pressure throughout the study period and undergo two additional study visits. At each study visit, participants will undergo a blood draw, blood pressure measurement and assessment of endothelial function with microiontophoresis. Participant adherence will be monitored through pill counts, text message check-ins, patient diary and biochemical monitoring.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, Investigators and outcomes assessors will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Group (Placebo Comparator): Similar appearing placebo pill daily for 6 months will be given to subjects.
  Interventions: Drug: Placebo
- Intervention Group (Experimental): Low-dose [81 mg] aspirin pill daily for 6 months will be given to subjects
  Interventions: Drug: Low-dose aspirin

INTERVENTIONS:
Drug: Low-dose aspirin — The intervention group will receive low-dose [81 mg] aspirin pill daily for 6 months.
  Arms: Intervention Group
Drug: Placebo — The control group will receive similar appearing placebo daily for 6 months.
  Arms: Placebo Group

SUMMARY:
The objective of this research project is to conduct a single-site pilot trial to assess the feasibility and effect of low-dose aspirin to augment vascular recovery in the immediate postpartum period after preeclampsia through two specific aims: 1) to pilot test the feasibility of conducting a randomized controlled trial of postpartum low dose aspirin vs. placebo, and 2) to assess the effect of postpartum aspirin on endothelial function and blood pressure. Our central hypothesis is that postpartum administration of low-dose aspirin following preeclampsia will be feasible, improve endothelial function, and lower BP at 6 months postpartum. Subjects will undergo 3 study visits involving BP measurements, blood draws, questionnaires, and/or microiontophoresis. Up to 60 adult subjects will be enrolled at Magee-Women's Hospital.

DETAILED DESCRIPTION:
This is a pilot randomized, single-center, double-blind placebo-control study of low dose aspirin in postpartum individuals with preeclampsia. Individuals will be randomized at the time of delivery 1:1 to 81mg of low-dose aspirin or identical appearing placebo daily for six months postpartum. Treatment and control groups will monitor home blood pressure throughout the study period and undergo two study visits. At each study visit, participants will undergo a blood draw, blood pressure measurement and assessment of endothelial function with microiontophoresis. Participant adherence will be monitored through pill counts, text message check-ins, patient diary and biochemical monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum individuals ≥18 years old
* Preeclampsia diagnosis

Exclusion Criteria:

* Fetal anomaly
* Multiple gestation
* Pre-pregnancy hypertension
* Allergy or contraindication to low-dose aspirin
* Pre-pregnancy diabetes

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent of participants eligible, enrolled and retained (feasibility) | Baseline to approximately 6 months postpartum
  To determine the feasibility of conducting a single-site randomized controlled trial of 6 months of postpartum low-dose aspirin vs. placebo in women with preeclampsia.

SECONDARY OUTCOMES:
Study visit systolic BP | 2 months postpartum
  Mean study visit systolic BP
Study visit diastolic BP | 2 months postpartum
  Mean study visit diastolic BP
Study visit systolic BP | 6 months postpartum
  Mean study visit systolic BP
Study visit diastolic BP | 6 months postpartum
  Mean study visit diastolic BP
Study visit mean arterial pressure | 2 months postpartum
  Mean study visit mean arterial pressure ((2*diastolic BP + systolic BP / 3))
Study visit mean arterial pressure | 6 months postpartum
  Mean study visit mean arterial pressure ((2*diastolic BP + systolic BP / 3))
Anti-hypertensive medication use | 2 months postpartum
  Use of anti-hypertensive medication (percent of participants)
Anti-hypertensive medication use | 6 months postpartum
  Use of anti-hypertensive medication (percent of participants)
Therapeutic intensity score | 2 months postpartum
  Therapeutic intensity score for those on anti-hypertensive medications. Range of scores 0 to 5 (higher number indicates higher doses and number of anti-hypertensive medications; worse outcome)
Therapeutic intensity score | 6 months postpartum
  Therapeutic intensity score for those on anti-hypertensive medications. Range of scores 0 to 5 (higher number indicates higher doses and number of anti-hypertensive medications; worse outcome)
Mean home systolic blood pressure | delivery through 6 months postpartum
  Mean home systolic blood pressure
Mean home diastolic blood pressure | delivery through 6 months postpartum
  Mean home diastolic blood pressure
Mean home mean arterial pressure | delivery through 6 months postpartum
  Mean home mean arterial pressure
Mean daytime systolic blood pressure | 6 months postpartum
  Mean daytime systolic blood pressure on ambulatory blood pressure monitoring
Mean nocturnal systolic blood pressure | 6 months postpartum
  Mean nocturnal systolic blood pressure on ambulatory blood pressure monitoring
Mean daytime diastolic blood pressure | 6 months postpartum
  Mean daytime diastolic blood pressure on ambulatory blood pressure monitoring
Mean nocturnal diastolic blood pressure | 6 months postpartum
  Mean nocturnal diastolic blood pressure on ambulatory blood pressure monitoring
Mean nocturnal mean arterial pressure | 6 months postpartum
  Mean nocturnal mean arterial pressure on ambulatory blood pressure monitoring
Mean daytime mean arterial pressure | 6 months postpartum
  Mean daytime mean arterial pressure on ambulatory blood pressure monitoring
Mean overall mean arterial pressure | 6 months postpartum
  Mean overall mean arterial pressure on ambulatory blood pressure monitoring
Mean overall systolic blood pressure | 6 months postpartum
  Mean overall systolic blood pressure on ambulatory blood pressure monitoring
Mean overall diastolic blood pressure | 6 months postpartum
  Mean overall diastolic blood pressure on ambulatory blood pressure monitoring
Classification of hypertension | 2 months postpartum
  Stage 1, stage 2 hypertension (percent of participants with each stage)
Classification of hypertension | 6 months postpartum
  Stage 1, stage 2 hypertension (percent of participants with each stage)
Endothelial function EC50% | 2 months postpartum
  EC50% from microiontophoresis
Endothelial function EC50% | 6 months postpartum
  EC50% from microiontophoresis
Endothelial function Emax | 2 months postpartum
  Emax from microiontophoresis
Endothelial function Emax | 6 months postpartum
  Emax from microiontophoresis
Endothelial function change in Emax | 2 to 6 months postpartum
  Change in Emax between visits
Endothelial function change in EC50% | 2 to 6 months postpartum
  Change in EC50% between visits
Change in systolic blood pressure | 2 to 6 months postpartum
  Change in study visit mean systolic blood pressure between visits
Change in diastolic blood pressure | 2 to 6 months postpartum
  Change in study visit mean diastolic blood pressure between visits
Change in mean arterial pressure | 2 to 6 months postpartum
  Change in study visit mean arterial pressure between visits

CONTACTS AND LOCATIONS:
Overall Officials: Alisse K Hauspurg, MD, Principal Investigator — UPMC Magee Women's Hospital
Locations (1):
- University of Pittsburgh Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data (including data dictionaries) will be shared at the discretion of the primary investigator. Data will include blood pressure, weight, demographics, physical activity, and pregnancy related information. Additional documents (such as the study protocol) will be made available.
Supporting Information: Study Protocol
Time Frame: Within a year after outcomes are published and no later than 3 years after the end of clinical activities.
Access Criteria: NHLBI data repository request process
URL: https://biolincc.nhlbi.nih.gov/home/